CLINICAL TRIAL: NCT03787784
Title: Automatic Classification of Colorectal Polyps Using Probe-based Endomicroscopy With Artificial Intelligence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2018SDU-QILU-8
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-09

CONDITIONS: Probe-based Confocal Laser Endomicroscopy; Artificial Intelligence; Colorectal Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI visible group (Experimental)
  Interventions: Other: AI presentation
- AI invisible group (No Intervention)

INTERVENTIONS:
Other: AI presentation — Automatic diagnosis information of AI is visible to endoscopist
  Arms: AI visible group

SUMMARY:
Probe-based confocal laser endomicroscopy (pCLE) is an endoscopic technique that enables real-time histological evaluation of gastrointestinal mucosa during ongoing endoscopy examination. It can predict the classification of Colorectal Polyps accurately. However this requires much experience, which limits the application of pCLE. The investigators designed a computer program using deep neural networks to differentiate hyperplastic from neoplastic polyps automatically in pCLE examination.

ELIGIBILITY:
Inclusion Criteria:

aged between 18 and 80; agree to give written informed consent.

Exclusion Criteria:

Patients under conditions unsuitable for performing CLE including coagulopathy , impaired renal or hepatic function, pregnancy or breastfeeding, and known allergy to fluorescein sodium; Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of classifying colorectal Polyps using Probe-based endomicroscopy with deep neural networks | 4 months
  The primary outcome is to test the diagnostic accuracy, sensitivity, specificity, PPV, NPV of the Artificial Intelligence for diagnosing Colorectal Polyps on real-time pCLE examination.

SECONDARY OUTCOMES:
Contrast the diagnosis efficiency of Artificial Intelligence with endoscopists | 3 month
  The secondary outcome is to compare the diagnosis efficiency (including diagnostic accuracy, sensitivity, specificity, PPV, NPV for diagnosing Colorectal Polyps on real-time pCLE examination) between Artificial Intelligence and endoscopists.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic unit of Qilu Hospital Shandong University, Jinan, Shandong, China